CLINICAL TRIAL: NCT01780480
Title: Dynamic Combination Therapy on Chinese Herbal Granules Based on Differentiation of Syndrome (Zhenghou)of Traditional Chinese Medicine to Improve the Symptoms in the Convalescent Phase of Ischemic Stroke: a Pilot Study
Brief Title: Dynamic Combination Therapy on Chinese Herbal Granules to Improve the Symptoms in Convalescent Phase of Ischemic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Zhong Wang, Professor, China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZYPF-201212
Record Dates: First submitted 2013-01-27; First posted 2013-01-31 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Ischemic Stroke; Convalescence
Keywords: Ischemic Stroke; Convalescence; Randomized Controlled Trial; Pilot Study; Traditional Chinese Medicine
MeSH Terms: conditions — Ischemic Stroke; Convalescence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dynamic Chinese herbal granule formula (Experimental): Based on standard medical care, after evaluated the style of the syndrome (Zhenghou) by an experienced integrative medicine doctor, the patients should be given a combination therapy of a Chinese herbal granule formula twice a day for 4 weeks, which should be selected from 10 kinds of Chinese herbal granules, including 3 gram of Huangqi(Astragalus root), 2 gram of Renshen(ginseng), 2.5 gram of Danggui(Angelica sinensis), 2 gram of Danshen(Salvia miltiorrhiza), 2 gram of Dilong(Geosaurus), 3 gram of Chishao(Radix Paeoniae Rubra), 2 gram of Honghua(Safflower), 2 gram of Chuanxiong(Rhizoma Chuanxiong), 2 gram of Sanqi(Radix Notoginseng), 3 gram of Shudihuang(Radix Rehmanniae Preparata). The Chinese herbal granule formula could be weekly changed according to differentiation of Zhenghou.
  Interventions: Drug: Dynamic Chinese herbal granule formula; Procedure: Standard medical care
- Placebo (Placebo Comparator): The process is the same as the experimental arm, except that the matched placebo granules should be in turn of Chinese herbal granules.
  Interventions: Drug: Placebo; Procedure: Standard medical care

INTERVENTIONS:
Drug: Dynamic Chinese herbal granule formula — After evaluated the style of the syndrome (Zhenghou) by an experienced integrative medicine doctor, the patients should be given a Chinese herbal granule formula twice a day for 4 weeks, which should be selected from 10 kinds of Chinese herbal granules and weekly changed according to differentiation of syndromes (Zhenghou) of patients.
  Arms: Dynamic Chinese herbal granule formula
Drug: Placebo — The 10 kinds of matched placebo granules were of the similar appearance, taste, smell with the corresponding Chinese herbal granules respectively. The interventional process of the placebo group is similar as the Chinese herbal granule formula group
  Arms: Placebo
Procedure: Standard medical care — Standard medical care is the basic treatment for all enrolled patients, including aspirin 75-100mg per day, standard rehabilitation training, treatment for their primary diseases, etc.

SUMMARY:
To evaluate the effect of the dynamic combination therapy on Chinese herbal granule formula (Fangji) based on differentiation of syndromes ("Zhenghou") according to the theory of traditional Chinese medicine for improving the symptoms in the convalescent phase of ischemic stroke, and to establish the pharmacodynamic model of "Zhenghou" according to the results of this trial.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 75 years.
* Clinical diagnosis of ischemic stroke causing a measurable neurological deficit defined as impairment of language, motor function, cognition and/or gaze, vision or neglect, confirmed by CT or MRI scan.
* Clinical diagnosis of "Qixu-Xueyu Zheng" (Qi deficiency and Blood Stasis Syndrome) as the scores of Chinese medicine symptoms scales in ischemic stroke on both "Qixue" and "Xueyu" ≥ 7.
* 15 days to 60 days after onset of symptoms.
* Clinical diagnosis of cerebral anterior circulation obstruction.
* 4≤NIHSS<20.
* Patient is willing to participate voluntarily and to sign a written patient informed consent.

Exclusion Criteria:

* Transient ischemic attack
* Evidence of intracranial hemorrhage (ICH) in 6 months
* Evidence of other cerebral diseases (eg.vascular malformation, tumor, abscess or multiple sclerosis etc.)on the CT or MRI scan.
* Woman with pregnancy, lactation or positive result of pregnancy test, or women who want to be pregnant in recent 6 months.
* Woman who is under menstrual period.
* Known history of allergy or suspected allergic to these chinese herbs.
* Complicated with atrial fibrillation.
* Fasting blood glucose ≥8 mmol / l under the treatment of diabetes or complicated with severe cardio-cerebrovascular diseases (eg. hyperlipemia, coronary heart disease with angina attack ≥ 4 times a day).
* Liver function impairment with the value of ALT or AST over 1.5-fold of normal value.
* Renal dysfunction with the value of serum creatinine over normal value.
* Prior disable patients or complicated with osteoarthropathy that influence the motor function of the limbs.
* With mental disorder that can not cooperate with doctor
* Suspected addicted into alcohol or drug abuse.
* With severe complications that would make the condition more complicated assessed by the investigator.
* Patient who is participating in other trials or has been participated in other trials in recent 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-01; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Symptom Scale of the "Qixu-Xueyu Zheng"(Qi Deficiency and Blood Stasis Syndrome) according to the theory of Traditional Chinese Medicine at Day 28 | Day 28

SECONDARY OUTCOMES:
Bathel Index | Day0; Day 7; Day 14; Day 21; Day 28; Day 90 after Onset
modified Rankin Scale | Day0; Day 7; Day 14; Day 21; Day 28; Day 90 after Onset
NIH stroke scale(NIHSS) | Day 0; Day7; Day 14; Day 21; Day 28; Day 90 after onset
EQ-5D scale | Day0; Day 7; Day 14; Day 21; Day 28; Day 90 after Onset
Overall mortality at day 90 | Day 90 after onset
Incidence of Recurrent Stroke | Day 90 after onset this time
Incidence of new-onset vascular events | Day 90 after onset this time
Incidence of adverse events (AEs) and serious AEs | From Day 0 to Day 90 after onset

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Wang, Dr., Study Chair — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences; Jun Liu, Dr., Principal Investigator — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences; Guang-qi Zhu, Study Director — The First Affiliated Hospital of Guiyang College of Traditional Chinese Medicine
Locations (1):
- The First Affiliated Hospital of Guiyang College of Traditional Chinese Medicine, Guiyang, Guizhou, China